CLINICAL TRIAL: NCT02736812
Title: Interest of Pre-hospital Administration of Lyophilized Plasma to Prevent or Treat Coagulopathy Associated With Post-traumatic Hemorrhagic Shock (PREHO-PLYO Study )
Brief Title: Pre-hospital Administration of Lyophilized Plasma for Post-traumatic Coagulopathy Treatment (PREHO-PLYO)
Acronym: PREHO-PLYO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Defence Health Service (Other Government)
Collaborators: Bataillon des marins pompiers de Marseille, France (Unknown); Military Hospital Laveran,Marseille, France (Unknown); Samu of Marseille, France (Unknown); Samu of Lyon, France (Unknown); Lyon-South Hospital, France (Unknown); Hôpital Edouard Herriot (Other); Fire Brigade Of Paris Emergency Medicine Dept (Other); CH Annecy Genevois (Other); Institut de Recherche Biomedicale des Armees (Other Government); Marseille North Hospital, France (Unknown); Samu of Necker, Paris, France (Unknown); Samu of Annecy, France (Unknown); Military Hospital Percy , Clamart, France (Unknown); Military Hospital Begin, Saint-Mandé, France (Unknown); Centre de transfusion sanguine des Armées, Clamart, France (Unknown); Henri Mondor University Hospital (Other); Samu of Beaujon, Clichy-La-Garenne, France (Unknown); Samu of Lariboisière, Paris, France (Unknown); Samu of Henri Mondor, Créteil, France (Unknown); Samu of Brest, Brest , France (Unknown); Samu of Pau , Pau , France (Unknown)
Responsible Party: Principal Investigator, Daniel Jost, Emergency Physician - Research Dept, Fire Brigade Of Paris Emergency Medicine Dept
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014RC04
Record Dates: First submitted 2016-03-27; First posted 2016-04-13 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Shock Hemorrhagic
Keywords: Randomized controlled trial; Lyophilized Plasma; Advanced Trauma Life Support Care
MeSH Terms: conditions — Shock, Hemorrhagic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- French Lyophilized Plasma (Experimental): receives French Lyophilized Plasma with the usual treatment for post traumatic hemorrhagic shock as given in the recommendations for best practice
  Interventions: Biological: French Lyophilized Plasma
- Normal Saline Solution (Active Comparator): receives Normale Saline Solution with the usual treatment of post traumatic hemorrhagic shock as given in the recommendations for best practice
  Interventions: Biological: Normale Saline Solution

INTERVENTIONS:
Biological: French Lyophilized Plasma — During the pre-hospital phase, the main events related to this arm are
  * Blood samples taken before treatment (TP, fibrinogen, platelets, RBC, grouping)
  * Usual pre-hospital care according to recommendations in best practices
  * Administration of FLYP
  Arms: French Lyophilized Plasma
Biological: Normale Saline Solution — During the pre-hospital phase, the main events related to this arm are
  * Blood samples taken before treatment (TP, fibrinogen, platelets, RBC, grouping)
  * Usual pre-hospital care according to recommendations in best practices
  * Administration of Normale Saline Solution
  Arms: Normal Saline Solution

SUMMARY:
In severe bleeding due to trauma, a decrease in coagulation factors maintains and promotes bleeding. The plasma allows, through its contribution of coagulation factors, early prevention or correction of this post-trauma induced coagulopathy. This study aims to measure the effectiveness of pre-hospital FLYP administration in case of traumatic hemorrhagic shock, in the occurrence or the treatment of a post traumatic induced coagulopathy.

Study Design

This is a randomized controlled multicenter open label study in two parallel groups.

Eligibility criteria : adult, victim of a hemorrhagic shock of traumatic origin with [systolic blood pressure <70 mmHg] or Shock Index >1.1 The patients will receive either FLYP either the usual treatment as given in the recommendations for best practice.

The primary endpoint is the International Normalized Ratio (INR) at hospital admission.

The study must confirm the link between causality of early administration of plasma in improving post-traumatic coagulopathy. The study must show safe usage in out-of-hospital situations and the ability of medical staff to meet the requirements of the health authorities in terms of product use as well as in terms of traceability of the victims and the treatment they received.

DETAILED DESCRIPTION:
In severe bleeding due to trauma, a fall in coagulation factors maintains and promotes bleeding. The plasma allows, through its contribution of coagulation factors, early prevention or correction of this post-traumatic coagulopathy.

This labile blood product has so far only been used in armed conflicts by military medical and surgical units deployed in External Operations (EXOP) to meet the logistical constraints of the operating environment and the need to have, without delay, therapeutic plasma to treat bleeding casualties. Unlike frozen plasma used in hospitals, FLYP is stored at room temperature and is reconstituted in less than 6 mins.

In the civilian world, FLYP could be used by health institutions who have major logistical difficulties which do not allow them to ensure a cold chain of sub-zero temperatures, or in extreme emergency situations with the need for an immediate therapeutic plasma supply. In this second indication, FLYP should be used until the fresh frozen plasma is thawed and available. Its use in pre-hospital situations is also justified due to its immediate availability and storage conditions.

FLYP is sterile and is in powder-form with a residual humidity not exceeding 2%. It is packaged in a sterile and pyrogenic glass vial.

The main objective is to measure the effectiveness of pre-hospital FLYP administration in case of traumatic hemorrhagic shock, in the occurrence or the treatment of a post traumatic coagulopathy.

The secondary objectives consist in assessing the following outcomes :

(1) the need for massive transfusion (3) the ICU length of stay (4) the survival rate on day 30 (5) FLYP prehospital usability in civilian population (the compilation of technical and logistical difficulties encountered with administration of FLYP) (6) the Prothrombin time (PT) at hospital admission. Normal values for PT are 70 - 130%.

(7) the fibrinogen level at hospital admission (8) the variation in the level of PT, between the pre-hospital setting and the hospital admission .

(9) the variation in the level of INR, between the pre-hospital setting and the hospital admission .

(10) the variation in the fibrinogen level between the pre-hospital setting and the hospital admission .

Method

The attribution of the experimental treatment (FLYP or saline), to each patient who will receive a treatment numbered from 1 to 140, was carried out in advance using STATA 14.0 software.

Type of randomisation : randomisation in blocks of 2, stratified by center.

Treatments are allocated to participants in each "pre-hospital" center by ascending number.

Participants and investigators are therefore not blinded to the allocated treatment.However, the statistical analysis is planned to be carried out as a blind study regarding knowledge of the allocated treatment.

The planned experimental design is identical for each pre-hospital investigation centre.

Care of a patient in traumatic hemorrhagic shock is identical from one investigating centre to another: it is based on formalized expert recommendations on hemorrhagic shock resuscitation.

Determination of the number of subjects required

Coagulation factors were measured in a pre-after study in 2010 in the army in severely traumatized patients. The "before" period consisted of an isotonic infusion of saline saline chlorine, the "after" period of FLYP transfusion. In total, the inclusion of 124 patients showed a significant difference between the two groups in terms of PT value. In the absence of any other data available at the time of writing the protocol, we have brought the number of subjects required to 140 (= 2X 70) according to a 10% in the follow-up.

There is no planned interim analysis.

The administration of the treatment in the study is stopped if any adverse event (AE) occurs (abnormal clinical manifestation,...) and the offending experimental treatment is retained. Usual care and corrective actions are continued in the field, during transport and at the receiving hospital. An independent oversight committee meeting is organized to discuss the stopping or the continuation of the study according to the nature of the AE.

Comparability of the 2 groups for the primary endpoint:

The median INR values are compared between the two groups, after adjustment on other variables if necessary.

Comparability of the 2 groups for the secondary endpoints:

* Transfusion requirement will be judged by the number of units transfused after arrival at the hospital: packed red blood cells (RBC), platelet concentrates, fibrinogen, coagulation factors and plasma. The transfusion requirement will be measured over a period of 24 to 48 hours.
* The median number of days in the ICU between the two groups will use the medians test
* Survival analysis up to 30 days will be based on the comparison of Kaplan-Meier curves, by the log-rank test, and a Cox model to estimate the role of administration of FLYP on survival, taking into account potential confounding factors.
* The usability of administering FLYP will be judged on the grounds of interruption or non-administration of the experimental treatment, depending on the ability to respect the procedure and the use of a Labile Blood Product according to the rules of good practice.
* The average differential (pre-hospital -hospital) of coagulation parameters between the two groups will be compared by an ANCOVA adjusted on other variables if needed.

INTERRUPTION OR STOPPING OF THE STUDY

The sponsor has the responsibility to report, to the national health authority , any serious and unexpected adverse events attributable to the labile blood product of cell therapy and/or protocol within 15 days (7 days in case of death and life-threatening situations).

In the case of occurrence of an incident, accident, or event, interruption of the study is planned after analysis and decision by the hemovigilance and safety committee of the study.

RISKS

A full report on the risks, the description of incidents, accidents and adverse events will be the subject of a chapter in the results section and also in the discussion.

FINANCING

Funding for the study is provided by the Health Department of the Army (promoter, following the acceptance of the study in the context of Clinical research projects in the Health service of armies).

DISCUSSION

The study must confirm the link between causality of early administration of plasma in improving post-traumatic coagulopathy.

The study must show safe usage in out-of-hospital situations and the ability of medical staff to meet the requirements of the health authorities in terms of product use as well as in terms of traceability of the victims and the treatment they received.

CONCLUSION

This is the first study that aims to assess the usability and efficiency of FLYP in prehospital situation.

ELIGIBILITY:
Inclusion Criteria:

* hemorrhagic shock of traumatic origin
* [Systolic Blood Pressure <70 mmHg] OR [Shock index > 1.1]

Exclusion Criteria:

* Refusal to participate in the research
* Unaffiliated to a social welfare system
* Age under 18 years
* Privation of person's liberty
* Person subject to a safeguard measure of justice
* Pregnancy
* Allergy known to Amotosalen® and psoralen
* Contribution factor clotting other than Plyo
* Patient initialy in cardiac arrest
* Patient initially in cardiac arrest, followed by resumption of spontaneous circulation
* People who could not have blood sample (required for the primary endpoint)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-04-01; Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
the International Normalized Ratio level (international unit IU) at hospital admission | 1 day

SECONDARY OUTCOMES:
number of plasma units administered at 24 and 48 hours | 48 hours
Number of RBC Concentrates units administered at 24 and 48 hours | 48 hours
Number of platelet concentrates units administered at 24 and 48 hours | 48 hours
Total Intensive care unit of stay (days) | 30 days
Survival | 30 days
FLYP prehospital usability in civilian population (questionnaire) | 30 days
  Compilation of technical and logistical difficulties encountered before, during and after administration of FLYP
Fibrinogen level (grams) | 1 day
Prothrombin level change (percentage) | 48 hours
  The difference in the level of Prothrombin (PT), between prehospital and hospital admission
the level of coagulation factors (international unit IU) at hospital admission | 1 day
Quantity of fibrinogen administered in grams at 24 and 48 hours | 48 hours
quantity of coagulation factors administered (international units IU) | 48 hours
  quantity of coagulation factors administered (international units IU)
Thromboelastometry median clotting time (CT) (minutes). | 1 hour
  Time in minutes and secondes for each step coming from rotational elastometry
Thromboelastometry median Clot Formation Time (CFT) in minutes and seconds | 1 hour
  Time in minutes and seconds for each step coming from rotational elastometry
Thromboelastometry median maximal lysis (ML) time in minutes ans seconds | 1 hour
  Time in minutes and seconds for each step coming from rotational elastometry
Thromboelastometry alpha angle (degrees) | 1 hour
  measure unit : degrees
Thromboelastometry median Maximal Clot Firmness (MCF) time in minutes and seconds | 1 hour
  Time in minutes and seconds for each step coming from rotational elastometry

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre TOURTIER, Professor, Study Chair — Fire Brigade Of Paris Emergency Medicine Dept; Daniel JOST, MD, Principal Investigator — Fire Brigade Of Paris Emergency Medicine Dept; Anne SAILLIOL, Professor, Study Chair — Centre de Transfusion Sanguine des Armées; Catherine VERRET, MD, Study Chair — Institut de recherche biomedicale des armées
Locations (22):
- France (22):
  - Centre Hospitalier Annecy Genevois, Annecy
  - Samu 74 Annecy Genevois, Annecy
  - Samu de BREST, Brest
  - Hopital d'instruction des Armées PERCY, Clamart
  - Centre de Transfusion Sanguine des Armées, Clamart
  - Hopital Beaujon, Clichy
  - Henri Mondor University Hospital, Créteil
  - Hopital Kremlin Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier EDOUARD HERRIOT, Lyon
  - Samu de LYON, Lyon
  - Centre Hospitalier LYON SUD, Lyon
  - Hopital d'Instruction des Armées LAVERAN, Marseille
  - Bataillon des marins-pompiers de Marseille, Marseille
  - Hopital Nord de Marseille, Marseille
  - Samu de Marseille, Marseille
  - Hopital Pitié Salpétrière, Paris
  - Hopital Europen Georges Pompidou, Paris
  - Samu de Paris, Paris
  - Fire Brigade Of Paris Emergency Medicine Dept, Paris
  - Smur Lariboisiere, Paris
  - Samu de PAU, Pau
  - Hopital des Instructions des Armées BEGIN, Saint-Mandé

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boutonnet M, Pasquier P, Salvadori A, Auroy Y, Tourtier JP. Advocacy to extend the use of continuous noninvasive hemoglobin measurement. Crit Care Med. 2011 Dec;39(12):2783-4; author reply 2784-5. doi: 10.1097/CCM.0b013e31822b3a22. No abstract available. PMID 22094519
- [Background] Pasquier P, Boutonnet M, Giraud N, Salvadori A, Tourtier JP. Hypotension redefined, shock index and massive transfusion. J Trauma. 2011 Sep;71(3):784-5. doi: 10.1097/TA.0b013e318228b83d. No abstract available. PMID 21909011
- [Background] Brohi K, Singh J, Heron M, Coats T. Acute traumatic coagulopathy. J Trauma. 2003 Jun;54(6):1127-30. doi: 10.1097/01.TA.0000069184.82147.06. PMID 12813333
- [Background] Martinaud C, Tourtier JP, Pasquier P, Ausset S, Sailliol A. The French freeze-dried plasma. J Trauma. 2011 Oct;71(4):1091-2. doi: 10.1097/TA.0b013e31822a8fd5. No abstract available. PMID 21986756
- [Background] Martinaud C, Ausset S, Deshayes AV, Cauet A, Demazeau N, Sailliol A. Use of freeze-dried plasma in French intensive care unit in Afghanistan. J Trauma. 2011 Dec;71(6):1761-4; discussion 1764-5. doi: 10.1097/TA.0b013e31822f1285. PMID 22182886
- [Background] Sailliol A, Martinaud C, Cap AP, Civadier C, Clavier B, Deshayes AV, Mendes AC, Pouget T, Demazeau N, Chueca M, Martelet FR, Ausset S. The evolving role of lyophilized plasma in remote damage control resuscitation in the French Armed Forces Health Service. Transfusion. 2013 Jan;53 Suppl 1:65S-71S. doi: 10.1111/trf.12038. PMID 23301975
- [Background] Martinaud C, Civadier C, Ausset S, Verret C, Deshayes AV, Sailliol A. In vitro hemostatic properties of French lyophilized plasma. Anesthesiology. 2012 Aug;117(2):339-46. doi: 10.1097/ALN.0b013e3182608cdd. PMID 22739764
- [Background] Glassberg E, Nadler R, Gendler S, Abramovich A, Spinella PC, Gerhardt RT, Holcomb JB, Kreiss Y. Freeze-dried plasma at the point of injury: from concept to doctrine. Shock. 2013 Dec;40(6):444-50. doi: 10.1097/SHK.0000000000000047. PMID 24089000
- [Background] Brown JB, Guyette FX, Neal MD, Claridge JA, Daley BJ, Harbrecht BG, Miller RS, Phelan HA, Adams PW, Early BJ, Peitzman AB, Billiar TR, Sperry JL. Taking the Blood Bank to the Field: The Design and Rationale of the Prehospital Air Medical Plasma (PAMPer) Trial. Prehosp Emerg Care. 2015 Jul-Sep;19(3):343-50. doi: 10.3109/10903127.2014.995851. Epub 2015 Feb 6. PMID 25658881
- [Background] Kim BD, Zielinski MD, Jenkins DH, Schiller HJ, Berns KS, Zietlow SP. The effects of prehospital plasma on patients with injury: a prehospital plasma resuscitation. J Trauma Acute Care Surg. 2012 Aug;73(2 Suppl 1):S49-53. doi: 10.1097/TA.0b013e31826060ff. PMID 22847094
- [Background] Chapman MP, Moore EE, Moore HB, Gonzalez E, Morton AP, Chandler J, Fleming CD, Ghasabyan A, Silliman CC, Banerjee A, Sauaia A. The "Death Diamond": Rapid thrombelastography identifies lethal hyperfibrinolysis. J Trauma Acute Care Surg. 2015 Dec;79(6):925-9. doi: 10.1097/TA.0000000000000871. PMID 26488324
- [Result] Floccard B, Rugeri L, Faure A, Saint Denis M, Boyle EM, Peguet O, Levrat A, Guillaume C, Marcotte G, Vulliez A, Hautin E, David JS, Negrier C, Allaouchiche B. Early coagulopathy in trauma patients: an on-scene and hospital admission study. Injury. 2012 Jan;43(1):26-32. doi: 10.1016/j.injury.2010.11.003. Epub 2010 Nov 26. PMID 21112053
- [Result] Borgman MA, Spinella PC, Perkins JG, Grathwohl KW, Repine T, Beekley AC, Sebesta J, Jenkins D, Wade CE, Holcomb JB. The ratio of blood products transfused affects mortality in patients receiving massive transfusions at a combat support hospital. J Trauma. 2007 Oct;63(4):805-13. doi: 10.1097/TA.0b013e3181271ba3. PMID 18090009
- [Result] de Biasi AR, Stansbury LG, Dutton RP, Stein DM, Scalea TM, Hess JR. Blood product use in trauma resuscitation: plasma deficit versus plasma ratio as predictors of mortality in trauma (CME). Transfusion. 2011 Sep;51(9):1925-32. doi: 10.1111/j.1537-2995.2010.03050.x. Epub 2011 Feb 18. PMID 21332727
- [Result] Peltan ID, Vande Vusse LK, Maier RV, Watkins TR. An International Normalized Ratio-Based Definition of Acute Traumatic Coagulopathy Is Associated With Mortality, Venous Thromboembolism, and Multiple Organ Failure After Injury. Crit Care Med. 2015 Jul;43(7):1429-38. doi: 10.1097/CCM.0000000000000981. PMID 25816119
- [Result] Holcomb JB, Tilley BC, Baraniuk S, Fox EE, Wade CE, Podbielski JM, del Junco DJ, Brasel KJ, Bulger EM, Callcut RA, Cohen MJ, Cotton BA, Fabian TC, Inaba K, Kerby JD, Muskat P, O'Keeffe T, Rizoli S, Robinson BR, Scalea TM, Schreiber MA, Stein DM, Weinberg JA, Callum JL, Hess JR, Matijevic N, Miller CN, Pittet JF, Hoyt DB, Pearson GD, Leroux B, van Belle G; PROPPR Study Group. Transfusion of plasma, platelets, and red blood cells in a 1:1:1 vs a 1:1:2 ratio and mortality in patients with severe trauma: the PROPPR randomized clinical trial. JAMA. 2015 Feb 3;313(5):471-82. doi: 10.1001/jama.2015.12. PMID 25647203
- [Result] Sunde GA, Vikenes B, Strandenes G, Flo KC, Hervig TA, Kristoffersen EK, Heltne JK. Freeze dried plasma and fresh red blood cells for civilian prehospital hemorrhagic shock resuscitation. J Trauma Acute Care Surg. 2015 Jun;78(6 Suppl 1):S26-30. doi: 10.1097/TA.0000000000000633. PMID 26002260
- [Result] Moore HB, Moore EE, Morton AP, Gonzalez E, Fragoso M, Chapman MP, Dzieciatkowska M, Hansen KC, Banerjee A, Sauaia A, Silliman CC. Shock-induced systemic hyperfibrinolysis is attenuated by plasma-first resuscitation. J Trauma Acute Care Surg. 2015 Dec;79(6):897-903; discussion 903-4. doi: 10.1097/TA.0000000000000792. PMID 26680132
- [Result] Rugeri L, Levrat A, David JS, Delecroix E, Floccard B, Gros A, Allaouchiche B, Negrier C. Diagnosis of early coagulation abnormalities in trauma patients by rotation thrombelastography. J Thromb Haemost. 2007 Feb;5(2):289-95. doi: 10.1111/j.1538-7836.2007.02319.x. Epub 2006 Nov 16. PMID 17109736
- [Derived] Brunskill SJ, Disegna A, Wong H, Fabes J, Desborough MJ, Doree C, Davenport R, Curry N, Stanworth SJ. Blood transfusion strategies for major bleeding in trauma. Cochrane Database Syst Rev. 2025 Apr 24;4(4):CD012635. doi: 10.1002/14651858.CD012635.pub2. PMID 40271704
- [Derived] Jost D, Lemoine S, Lemoine F, Derkenne C, Beaume S, Lanoe V, Maurin O, Louis-Delauriere E, Delacote M, Dang-Minh P, Franchin-Frattini M, Bihannic R, Savary D, Levrat A, Baudouin C, Trichereau J, Salome M, Frattini B, Ha VHT, Jouffroy R, Seguineau E, Titreville R, Roquet F, Stibbe O, Vivien B, Verret C, Bignand M, Travers S, Martinaud C, Arock M, Raux M, Prunet B, Ausset S, Sailliol A, Tourtier JP; Prehospital Lyophilized Plasma (PREHO-PLYO) Study Group. Prehospital Lyophilized Plasma Transfusion for Trauma-Induced Coagulopathy in Patients at Risk for Hemorrhagic Shock: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2223619. doi: 10.1001/jamanetworkopen.2022.23619. PMID 35881397
- [Derived] Jost D, Lemoine S, Lemoine F, Lanoe V, Maurin O, Derkenne C, Franchin Frattini M, Delacote M, Seguineau E, Godefroy A, Hervault N, Delhaye L, Pouliquen N, Louis-Delauriere E, Trichereau J, Roquet F, Salome M, Verret C, Bihannic R, Jouffroy R, Frattini B, Hong Tuan Ha V, Dang-Minh P, Travers S, Bignand M, Martinaud C, Garrabe E, Ausset S, Prunet B, Sailliol A, Tourtier JP; PREHO-PLYO Study Group. French lyophilized plasma versus normal saline for post-traumatic coagulopathy prevention and correction: PREHO-PLYO protocol for a multicenter randomized controlled clinical trial. Trials. 2020 Jan 22;21(1):106. doi: 10.1186/s13063-020-4049-1. PMID 31969168